CLINICAL TRIAL: NCT05861141
Title: Effect of Aerobic Training on Sleep Problems and Pulmonary Functions in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mayar Abdel Mohsen Ahmed Magd Behairy, Physiotherapy Practitioner, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004243
Record Dates: First submitted 2023-04-05; First posted 2023-05-16 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Down Syndrome
Keywords: Aerobic Training; Treadmill Training; Sleep; Sleep Problems; Sleep Disturbances; Obstructive Sleep Apnea (OSA); Pulmonary Functions; Down Syndrome; Trisomy 21; Children's Sleep Habits Questionnaire (CSHQ); Handheld Spirometer
MeSH Terms: conditions — Down Syndrome; Parasomnias; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Patients will receive a selected physical therapy program only.
  Interventions: Other: Selected physical therapy program
- Study Group (Experimental): Patients will receive the same selected physical therapy program as the control group in addition to aerobic exercise in the form of treadmill training.
  Interventions: Device: Aerobic training

INTERVENTIONS:
Other: Selected physical therapy program — Patients will receive a selected physical therapy program for 1 hr, 3 times per week, for 3 successive months in the form of:
  * Balance and postural control exercises for 15 minutes, including the following:
    * Standing on balance board.
    * Stoop and recovery.
  * Gait training for 45 minutes, including the following:
    * Forward, backward, and sideways walking.
    * Walking with obstacles using wedges and rolls with different diameters and heights.
  Arms: Control Group
Device: Aerobic training — Patients will receive the same selected physical therapy program as the control group for 15 minutes in addition to treadmill training for 45 minutes, 3 times per week, for 3 successive months.
  Treadmill training: Will be practiced according to the following stages:
  A- Warm up: 5 minutes.
  B- The exercise phase: 35 minutes (three-minute stages), the speed will be increased gradually every 3 minutes intervals until the child no longer be able to walk at the current stage.
  C- Cool down: 5 minutes.
  Other Names: Treadmill training
  Arms: Study Group

SUMMARY:
The study will be conducted to determine the effect of aerobic training on sleep problems and pulmonary functions in children with Down syndrome.

DETAILED DESCRIPTION:
The study will be carried out on 30 children with Down syndrome (trisomy 21) of both sexes, with ages ranging from 7 to 12 years old. Children will be recruited from schools for children with special needs. Children will be randomly assigned into two equal groups (control and study groups), 15 for each group. The control group will receive a selected physical therapy program only, while the study group will receive the same selected physical therapy program as the control group in addition to aerobic exercise in the form of treadmill training. The Arabic version of the Children's Sleep Habits Questionnaire (CSHQ) will be used to assess sleep problems, while a handheld spirometer will be used to assess pulmonary functions (forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), FEV1/FVC ratio, and peak expiratory flow rate (PEFR)) pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children with Down syndrome (trisomy 21).
* Their ages range from 7 to 12 years old.
* Both sexes will be included.
* Children should be able to understand and follow simple verbal commands or instructions (intelligence quotient (IQ) range: 50-70).
* Children should be able to walk independently.
* Their total scores on the Arabic version of the Children's Sleep Habits Questionnaire (CSHQ) equal 41 or higher.

Exclusion Criteria:

Children will be excluded from the study if they:

* Have visual or hearing defects.
* Have spinal abnormality such as kyphosis and scoliosis.
* Have history of pulmonary infection and surgery of thoracic and abdominal region within the past 6 months.
* Play any specific sport or exercises.
* Have physical activity restrictions.
* Have musculoskeletal disorder.
* Take medications known to affect sleep.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Sleep Problems: | 6 months
  Will be measured by the Arabic version of the Children's Sleep Habits Questionnaire (CSHQ):
  A 33-item retrospective parent-report questionnaire was created as a screening tool for sleep issues over a "typical" recent week. Each item is scored 1-3 (1 = Rarely, 0-1x/week; 2 = Sometimes, 2-4x/week; 3 = Usually, 5-7x/week). There are 6 questions with reverse scoring in order to consistently make a higher score indicative of more disrupted sleep. This will yield a total score between 33 and 99. A total score of 41 or higher suggests the presence of a sleep disturbance.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC): | 6 months
  Pulmonary Functions:
  FVC will be measured by a handheld spirometer.
Forced Expiratory Volume in 1 second (FEV1): | 6 months
  Pulmonary Functions:
  FEV1 will be measured by a handheld spirometer.
FEV1/FVC ratio: | 6 months
  Pulmonary Functions:
  FEV1/FVC ratio will be measured by a handheld spirometer.
Peak Expiratory Flow Rate (PEFR): | 6 months
  Pulmonary Functions:
  PEFR will be measured by a handheld spirometer.

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa A Zaky, PhD, Principal Investigator — Professor of Physical Therapy for Pediatrics, Faculty of Physical Therapy, Cairo University; Saly S Abd Elhady, PhD, Principal Investigator — Lecturer of Physical Therapy for Pediatrics, Faculty of Physical Therapy, Cairo University
Locations (1):
- Cairo University, Cairo, Egypt